CLINICAL TRIAL: NCT00208143
Title: Seroquel (Quetiapine) Therapy for Schizophrenia and Schizoaffective Disorders and Comorbid Cocaine and/or Amphetamine Abuse/Dependence: A Comparative Study With Risperidone
Brief Title: Seroquel Therapy for Substance Use Disorders Comorbid With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Syed P. Sattar, M.D., Creighton University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRUSQUET00292
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2006-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Substance Abuse; Substance Dependence
Keywords: Cocaine Abuse; Cocaine Dependence; Amphetamine Abuse; Amphetamine Dependence; Schizophrenia; Comorbid; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Cocaine-Related Disorders; Amphetamine-Related Disorders | interventions — Quetiapine Fumarate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine
Drug: Risperidone

SUMMARY:
It is hypothesized that the atypical antipsychotic, Seroquel, will cause significant reduction in drug and alcohol cravings in patients with schizophrenia and comorbid cocaine and/methamphetamine dependence compared to the atypical antipsychotic, risperidone (Risperdal).

Patients treated with Seroquel will have less use of cocaine and/or methamphetamine as measured by the Time Line Follow-back, over a 24-week follow-up period.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental illness that afflicts approximately 1% of the population (1). Often these patients have comorbid cocaine and amphetamine dependence, which increases the severity of psychotic symptoms associated with schizophrenia, decreases treatment compliance and worsens prognosis.

The treatment of schizophrenia with comorbid cocaine and/or amphetamine dependence is complex and involves adherence to psychiatric medications, most often antipsychotic agents, along with participation in specific substance abuse treatment such as structured living, attendance at self-help group meetings, individual and group therapy and a commitment to sobriety. In the absence of specific pharmacotherapy of cocaine and amphetamine dependence, various antipsychotic medications have been compared to see if they impact comorbid cocaine and amphetamine abuse in addition to their antipsychotic effects.

The primary objective of this study is to test whether Seroquel as a mono-therapy decreases cocaine and/or methamphetamine use in patients with schizophrenia as compared to risperidone.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 19 - 65.
2. Diagnosis of schizophrenia or schizoaffective disorder with comorbid cocaine and/or amphetamine abuse/dependence as confirmed by Structured Clinical Interview for DSM-IV.
3. Comorbid diagnoses of depression, anxiety and/or personality disorders are permitted.
4. Ability to provide signed informed consent.
5. Stable general medical health.

Exclusion Criteria:

1. Dangerous to self or others.
2. Pregnancy, inability or unwillingness to use approved methods of birth control.
3. Inability or unwillingness to provide signed informed consent.
4. Diagnosis of bipolar disorder, primary major depressive disorder (As major Axis I diagnosis).
5. Inability to attend outpatient research clinic.
6. Medical conditions, which would preclude use of Seroquel.
7. Absolute need for ongoing treatment with antipsychotic other than Seroquel.
8. Medical instability defined as likelihood of needing to change prescription medication during the course of the study.
9. Patients currently taking quetiapine or risperidone.
10. Patients with unsuccessful treatment with quetiapine or risperidone.
11. Subjects with a HAM-D score of ≥20 at screening.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-11; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
50% or greater decrease in the drug use determined by the Time Line Follow Back method versus baseline.

SECONDARY OUTCOMES:
Psychiatric symptoms will be assessed with the CGI, PANSS, BPRS, HAM-D, and HAM-A.Safety and tolerability will be assessed by patient and physician reported adverse events and AIMS.Quality of life will be assessed with QoLI.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Petty, MD, PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Psychiatry and Research Center, Omaha, Nebraska, United States